CLINICAL TRIAL: NCT03132610
Title: Efficacy and Safety of Combined With Andrographolide Sulfonate on the Basis of Conventional Therapy in Patients With Acute Exacerbation of Chronic Bronchitis: a Randomized, Single Blind, Placebo-controlled, Multicenter Study
Brief Title: A Study of Andrographolide Sulfonate in Patients With Acute Exacerbation of Chronic Bronchitis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangxi Qingfeng Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JXQF-XYP-1608
Record Dates: First submitted 2017-04-13; First posted 2017-04-28 (Actual); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Acute Exacerbation of Chronic Bronchitis
MeSH Terms: interventions — andrographolide sulfonate

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Experimental group (Active Comparator): Conventional Therapy + Xiyanping injection(andrographolide sulfonate)
  Interventions: Drug: andrographolide sulfonate
- control group (Placebo Comparator): Conventional Therapy + Xiyanping injection simulation/andrographolide sulfonate simulation(0.9% normal saline)
  Interventions: Drug: andrographolide sulfonate simulation

INTERVENTIONS:
Drug: andrographolide sulfonate — Conventional Therapy+Xiyanping injection
  Other Names: Xiyanping injection
  Arms: Experimental group
Drug: andrographolide sulfonate simulation — Conventional Therapy+Xiyanping injection simulation
  Other Names: Xiyanping injection simulation
  Arms: control group

SUMMARY:
A multicenter,randomized,single-blind, placebo-controlled,phase 4 clinical trial to evaluate the efficacy and safety of andrographolide sulfonate in patients with acute exacerbation of chronic bronchitis

DETAILED DESCRIPTION:
The patient after passing the screening, with the ratio of 1:1, were randomly assigned to experimental group or control group. Experimental group: on the basis of Conventional Therapy,Xiyanping injection(andrographolide sulfonate) 10-20ml/d, With 0.9% normal saline 100ml-250ml diluted intravenous drip (not with other drugs in the same container mixed use), control drip speed per minute of 30-40 drops. control group: on the basis of Conventional Therapy,Xiyanping injection simulation(0.9% normal saline) 10-20ml/d, The treatment method is the same as the experimental group.

ELIGIBILITY:
Inclusion Criteria:

* 1.18-75 years, males or females;
* 2.patients met the acute exacerbation of chronic bronchitis diagnosis;
* 3.Patients with bronchitis were acute attacked 2-6 days,who had a history of chronic bronchitis more than 2 years.
* 4. Patients compliance is good, written informed consent was obtained from all participants before the study.

Exclusion Criteria:

* 1.Patients had a history of andrographolide sulfonate or andrographolide allergy.
* 2.Pregnancy, lactation, and absence of contraception in women of fertile age.
* 3.Judging by the researchers, Past or present illness of patients may affect to participate in the trial or affect the outcome of the study, including cardio-pulmonary diseases, malignant diseases, autoimmune diseases, hepatorenal disease, blood diseases, nervous system diseases, immune system diseases and endocrine diseases
* 4.After checking, Patients with pulmonary tuberculosis, bronchial asthma, bronchial pneumonia, bronchiectasis, pneumoconiosis, silicosis, lung cancer, pulmonary infiltration or other allergic respiratory diseases and other chronic lung diseases
* 5.Patients using systemic steroids or other immunosuppressive therapy
* 6.Patients with severe cardiopulmonary dysfunction, abnormal liver and kidney function, blood system diseases
* 7.Patients are alcohol (daily drink alcoholic wine is more than 40g) or drug abuse or drug addicts in the past year.
* 8.Patients were participated in any study of drug trials in the last 30 days.
* 9.According to the researchers' judgment, anyone who are not suitable for the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2016-12-01 (Actual); Primary Completion 2017-12-01 (Estimated); Study Completion 2018-06-01 (Estimated)

PRIMARY OUTCOMES:
cured rate | less than 14 days
  clinical symptoms(fever, cough, expectoration and gasp) and signs totally disappear, the period of lab tests（WBC,CRP, chest X-ray） return to normal is recorded。

SECONDARY OUTCOMES:
effective time window | less than 14 days
  days range from treatment is received to the effectiveness is observed, and symptoms disappear (fever, cough, expectoration and gasp).
days of antibiotic use | less than 14 days
  oral anti infective drugs use days and intravenous anti infective drugs use days are recorded
the incidence of complications | less than 14 days
  such as, the incidence of Acute otitis media, acute rhinitis, acute bronchitis, acute bronchitis, and so on.
bacterial eradication rate | less than 14 days
  bacterial eradication rate=Sputum culture negative cases after treatment /sputum culture positive cases before treatment x 100%
  =Sputum culture negative cases after treatment /sputum culture positive cases before treatment x 100%
direct medical cost | less than 14 days
  medical cost including hospital expenses, examine fee, medication fee, et al, relate to treatment in hospital
number of participants with treatment-related adverse events | less than 14 days
  the total incidence of adverse events, the incidence of adverse events associated with Xiyanping injection, the incidence of patients with grade 3 through grade 4 adverse events that are related to study drug, graded according to NCI-CTC V4.0 .
  Observe and record all adverse events and serious adverse events, including physical examination, vital signs, laboratory tests (Hematology, blood biochemistry, urine routine, stool routine), ECG changes and so on.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Zhang, Principal Investigator — The First Affiliated Hospital of Nanchang University; Ping Xu, Principal Investigator — The Fourth Affiliated Hospital of Nanchang University
Locations (1):
- The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi, China

IPD SHARING:
Plan to Share IPD: Undecided